CLINICAL TRIAL: NCT03347669
Title: A Pilot Study of Small Fiber Neuropathy Prevalence in Fibromyalgia Patients Compared to Healthy Subjects Using Sudoscan®
Acronym: NEFI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-362
Record Dates: First submitted 2017-11-08; First posted 2017-11-20 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Small fiber neuropathy; Sudoscan®
MeSH Terms: conditions — Fibromyalgia; Small Fiber Neuropathy

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FM patients (Experimental): 50 fibromyalgia patients/50 healthy subjects
  Interventions: Device: Sudoscan®
- Healthy subjects (Active Comparator): 50 fibromyalgia patients/50 healthy subjects
  Interventions: Device: Sudoscan®

INTERVENTIONS:
Device: Sudoscan® — Sudoscan® is a new device that provides rapid, non-invasive and reproducible quantitative assessment of sweat function. It makes it possible to measure the ability of the sweat glands to release chloride ions in response to electrochemical activation and thus to detect the presence of a neuropathy with small fibers. This new device therefore makes it possible to detect an SFN in a much simpler and faster way than the technique of ophthalmology, or biopsy. Sudoscan® has been tested to assess the neuropathies of small nerve fibers in several diseases, in particular diabetes, chemotherapy-induced polyneuropathy, familial amyloid polyneuropathy or Fabry disease. The interest of Sudoscan® lies in the fact that this device is non-invasive and rapid. Its diagnostic value has been compared with other neurophysiological tests.

SUMMARY:
Fibromyalgia (FM) is characterized by chronic diffuse pain and affects 0.5 to 5% of the population, with a higher prevalence in women1. This condition is characterized by joint and muscle pain, also associated with fatigue, migraine, sleeps disorders, depression and irritable bowel syndrome2. The presentation of these various symptoms varies greatly from one patient to another, with great heterogeneity in clinical, physical, social, psychological and therapeutic responses. . A recent parliamentary inquiry report called for recognition of the disease and recommended to build a unified care path for patients; a collective expertise is led by INSERM to help in patient care. Faced with the heterogeneity of FM, several international studies have attempted to identify subgroups of patients based essentially on clinical symptoms of the disease3-8, including a recent Korean study of 313 patients9, which suggested four groups, but with methodological limitations, not taking into account the new criteria10 for evaluating FM.

Recent studies have also shown that there is a peripheral neuropathic component in the mechanisms of this pathology, demonstrated by a decrease in the density of the epidermal nerve fibers11-12, called small fiber neuropathy (SFN) neuropathy. It is an attack of small sensory and sympathetic nerve fibers, causing pain, paresthesia as well as disturbances of the autonomous system. Other studies also suggested that a significant proportion of patients diagnosed with fibromyalgia had SFN, demonstrated by cutaneous biopsy13-14 or confocal microscopy of the cornea15. A new device, the Sudoscan®, makes it possible to detect a SFN much simpler, faster and less invasive than the technique of ophthalmology or biopsy. Although this Sudoscan® test has been used extensively in conditions such as diabetes16-19, no study has been used to assess the presence of SFN in FM.

The aim of this pilot study is to identify the prevalence of SFN in FM patients, using this new non-invasive device, in order to have a better defined representation of the prevalence of small-fiber neuropathy in an FM population compared to a group of healthy volunteer matched in age, sex, BMI and by menopausal status for women.

DETAILED DESCRIPTION:
Only one visit (2 to 3h) :

Inclusion of the patient Clinical examination ; evaluation of pain for FM patients Measurement of the electrochemical conductance of the hands and feet using Sudoscan® Evaluation of quality of life, anxiety, depression, sleep quality, fatigue, catastrophizing and social precarity End of study

ELIGIBILITY:
Inclusion Criteria:

* - Patient over 18 years of age and under 65 years of age,
* Male or female patient,
* Patient with fibromyalgia (according to the ACR criteria of 2016),
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Acceptance of written consent,
* Affiliation to the French Social Security system.

Inclusion criteria healthy subjects:

* Subject of more than 18 years,
* Woman or man,
* Healthy voluntary non-painful subjects matched by age (+/- 5 years), by sex, by BMI (+/- 10%) and by menopausal status for women,
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Acceptance of written consent,
* Affiliation to the French Social Security system,
* Registration or acceptance of registration in the National Register of Volunteers participating in research.

Exclusion Criteria:

* Exclusion criteria patients:
* Patient with a physical inability to place the palms of the hands or the soles of the feet on the electrodes of Sudoscan®,
* Patient with a medical and / or surgical history judged by the investigator or his representative to be incompatible with the test (in particular a disease known to give neuropathies of small fibers: diabetes, Gougerot-Sjögren's disease, vasculitis, sarcoidosis, chronic ethylism ...),
* Pregnant or nursing woman
* Patient participating in another clinical trial, or in a period of exclusion, or having received a total amount of compensation in excess of EUR 4500 over the 12 months preceding the start of the trial,
* Patient benefiting from a measure of legal protection (curatorship, guardianship, safeguard of justice ...),
* Patient not affiliated to the French Social Security system.

Exclusion criteria healthy subjects :

* Physical inability to place the palms of the hands or the soles of the feet on the electrodes of Sudoscan®.
* Medical and / or surgical history judged by the investigator or his representative to be incompatible with the test,
* Pregnant or nursing woman
* Participating in another clinical trial, or within the exclusion period, or having received a total amount of compensation in excess of EUR 4500 over the 12 months preceding the start of the trial,
* Cooperation and an understanding that does not permit strict compliance with the conditions laid down in the Protocol,
* Benefiting from a measure of legal protection (curatorship, guardianship, safeguard of justice ...),
* Not affiliated to the French Social Security system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Measure of the electrochemical conductance (µS) using Sudoscan® | at day 1
  Evaluation of the prevalence of fibromyalgia patients with small fibro neuropathy in comparison with healthy volunteers by measuring the electrochemical conductance of the palms of the hands (middle right and left hands) and feet (middle right and left) in μS using Sudoscan®.

SECONDARY OUTCOMES:
Biometric criteria | at day 1
  Collection of the age in years
Biometric criteria | at day 1
  Collection of sex, (male or female)
Biometric criteria | at day 1
  Collection weight in kilograms, height in meters, weight and eight will be combined to report BMI in kg/m²,
Biometric criteria | at day 1
  phototype Fitzpatrick classification
Numerical scale | at day 1
  This scale allows the patient to note pain on a graduation with a minimum score of 0 and a maximum score of 10. Higher value represent worse outcome.
Brief Pain Inventory | at day 1
  The BPI gives two main scores: a pain severity score and a pain interference score
Fibromyalgia Impact Questionnaire | at day 1
  The revised FIQ questionnaire is a 10-item self-questionnaire that assesses the impact of fibromyalgia. The first item is subdivided into 10 questions that assess the impact of the disease in everyday life
Quality of life (SF-12) | at day 1
  12 questions and an index is determined for both physical and mental health (0-100). Higher scores indicate greater physical and mental health
Anxiety and Depression (HAD) | at day 1
  The HAD scale is a 14-item self-administered questionnaire completed by the patient. These items are divided into two subscales: 7 items to assess depression and 7 items to assess anxiety. Higher value represent worse outcome.
Depression (Beck Depression Inventory) | at day 1
  Each item consists of 4 sentences corresponding to 4 degrees of increasing intensity of a symptom: from 0 to 3. In the counting, it is necessary to take into account the highest rating chosen for the same series. The overall score is obtained by adding the scores of the 13 items. The range of the scale is from 0 to 39. The higher the score, the more the subject is depressed.
Pittsburgh Sleep Quality Index | at day 1
  19-item self-administered questionnaire used to assess the quality of sleep. Higher value represent worse quality of sleep.
Chronic fatigue Severity Scale | at day 1
  9-item self-questionnaire to assess the patient's fatigue intensity. The patient is asked to circle a number from 1 to 7 for each question, a low value representing a low intensity. Higher value represents worse fatigue.
Pain Catastrophizing Scale | at day 1
  This questionnaire consists of 13 items. The patient will have to indicate how much he has thoughts or emotions when he feels pain by giving a score between 0 and 4, 0: not at all, 4: all the time. The final score is the sum of the scores for each question. Higher value represent worse outcome.
Assessment of socio-professional category, precariousness and health inequalities (Score EPICES). | at day 1
  The EPICES questionnaire consists of 11 binary questions (yes / no) to calculate an individual score indicating the precariousness and inequalities of health ranging from 0 to 100. Higher value represent worse outcome.
Measure of the electrochemical conductance (µS) using Sudoscan® | at day 1
  Assess the reproducibility (2 passes) of Sudoscan® in each participant: measurement of the electrochemical conductance of the palms of the hands (middle right and left hands) and feet (middle right and left) in μS using the Sudoscan®, 30 minutes after the first measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Perrot S, Choy E, Petersel D, Ginovker A, Kramer E. Survey of physician experiences and perceptions about the diagnosis and treatment of fibromyalgia. BMC Health Serv Res. 2012 Oct 10;12:356. doi: 10.1186/1472-6963-12-356. PMID 23051101
- [Background] Tagami J, Tao L, Pashley DH. Correlation among dentin depth, permeability, and bond strength of adhesive resins. Dent Mater. 1990 Jan;6(1):45-50. doi: 10.1016/0109-5641(90)90044-f. PMID 2198182
- [Background] Aktas A, Walsh D, Rybicki L. Symptom clusters: myth or reality? Palliat Med. 2010 Jun;24(4):373-85. doi: 10.1177/0269216310367842. PMID 20507866
- [Background] Flor H, Turk DC. Psychophysiology of chronic pain: do chronic pain patients exhibit symptom-specific psychophysiological responses? Psychol Bull. 1989 Mar;105(2):215-59. doi: 10.1037/0033-2909.105.2.215. PMID 2648442
- [Background] Giesecke T, Williams DA, Harris RE, Cupps TR, Tian X, Tian TX, Gracely RH, Clauw DJ. Subgrouping of fibromyalgia patients on the basis of pressure-pain thresholds and psychological factors. Arthritis Rheum. 2003 Oct;48(10):2916-22. doi: 10.1002/art.11272. PMID 14558098
- [Background] Wilson HD, Robinson JP, Turk DC. Toward the identification of symptom patterns in people with fibromyalgia. Arthritis Rheum. 2009 Apr 15;61(4):527-34. doi: 10.1002/art.24163. PMID 19333980
- [Background] de Souza JB, Goffaux P, Julien N, Potvin S, Charest J, Marchand S. Fibromyalgia subgroups: profiling distinct subgroups using the Fibromyalgia Impact Questionnaire. A preliminary study. Rheumatol Int. 2009 Mar;29(5):509-15. doi: 10.1007/s00296-008-0722-5. Epub 2008 Sep 27. PMID 18820930
- [Background] Bergman S. Psychosocial aspects of chronic widespread pain and fibromyalgia. Disabil Rehabil. 2005 Jun 17;27(12):675-83. doi: 10.1080/09638280400009030. PMID 16012060
- [Background] Salaffi F, Mozzani F, Draghessi A, Atzeni F, Catellani R, Ciapetti A, Di Carlo M, Sarzi-Puttini P. Identifying the symptom and functional domains in patients with fibromyalgia: results of a cross-sectional Internet-based survey in Italy. J Pain Res. 2016 May 13;9:279-86. doi: 10.2147/JPR.S100829. eCollection 2016. PMID 27257392
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Caro XJ, Winter EF. Evidence of abnormal epidermal nerve fiber density in fibromyalgia: clinical and immunologic implications. Arthritis Rheumatol. 2014 Jul;66(7):1945-54. doi: 10.1002/art.38662. PMID 24719395
- [Background] Doppler K, Rittner HL, Deckart M, Sommer C. Reduced dermal nerve fiber diameter in skin biopsies of patients with fibromyalgia. Pain. 2015 Nov;156(11):2319-2325. doi: 10.1097/j.pain.0000000000000285. PMID 26164586
- [Background] Oaklander AL, Herzog ZD, Downs HM, Klein MM. Objective evidence that small-fiber polyneuropathy underlies some illnesses currently labeled as fibromyalgia. Pain. 2013 Nov;154(11):2310-2316. doi: 10.1016/j.pain.2013.06.001. Epub 2013 Jun 5. PMID 23748113
- [Background] Uceyler N, Zeller D, Kahn AK, Kewenig S, Kittel-Schneider S, Schmid A, Casanova-Molla J, Reiners K, Sommer C. Small fibre pathology in patients with fibromyalgia syndrome. Brain. 2013 Jun;136(Pt 6):1857-67. doi: 10.1093/brain/awt053. Epub 2013 Mar 9. PMID 23474848
- [Background] Ramirez M, Martinez-Martinez LA, Hernandez-Quintela E, Velazco-Casapia J, Vargas A, Martinez-Lavin M. Small fiber neuropathy in women with fibromyalgia. An in vivo assessment using corneal confocal bio-microscopy. Semin Arthritis Rheum. 2015 Oct;45(2):214-9. doi: 10.1016/j.semarthrit.2015.03.003. Epub 2015 Mar 19. PMID 26094164
- [Background] Karnaukhov VK. [Significance of dyskinesia of the large intestine in the diagnosis of nonspecific ulcerative colitis]. Sov Med. 1973 Apr;36(4):97-100. No abstract available. Russian. PMID 4770015
- [Background] Selvarajah D, Cash T, Davies J, Sankar A, Rao G, Grieg M, Pallai S, Gandhi R, Wilkinson ID, Tesfaye S. SUDOSCAN: A Simple, Rapid, and Objective Method with Potential for Screening for Diabetic Peripheral Neuropathy. PLoS One. 2015 Oct 12;10(10):e0138224. doi: 10.1371/journal.pone.0138224. eCollection 2015. PMID 26457582
- [Background] Agarwal R, Gupta KP, Kumar S, Mehrotra NK. Assessment of some tumorigenic risks associated with fresh and used cutting oil. Indian J Exp Biol. 1986 Aug;24(8):508-10. No abstract available. PMID 3817891
- [Background] Mao F, Liu S, Qiao X, Zheng H, Xiong Q, Wen J, Liu L, Tang M, Zhang S, Zhang Z, Ye H, Lu B, Li Y. Sudoscan is an effective screening method for asymptomatic diabetic neuropathy in Chinese type 2 diabetes mellitus patients. J Diabetes Investig. 2017 May;8(3):363-368. doi: 10.1111/jdi.12575. Epub 2016 Oct 5. PMID 27607763
- [Derived] Pickering G, Achard A, Corriger A, Sickout-Arondo S, Macian N, Leray V, Lucchini C, Cardot JM, Pereira B. Electrochemical Skin Conductance and Quantitative Sensory Testing on Fibromyalgia. Pain Pract. 2020 Apr;20(4):348-356. doi: 10.1111/papr.12857. Epub 2019 Dec 24. PMID 31705738